CLINICAL TRIAL: NCT05873127
Title: A Randomized Controlled Study of Web-based Guided Self-help CBT-E Versus Online Group CBT-E for Binge Eating Behavior
Brief Title: Web-based Guided Self-help CBT-E vs Online G-CBT-E for Binge Eating Behavior
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202140092
Record Dates: First submitted 2023-04-23; First posted 2023-05-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- web-based guided self-help CBT-E (Experimental): After randomization, 8-10 patients were assigned to self-help CBT-E group each time.
  Interventions: Behavioral: web-based guided self-help Enhanced Cognitive Behavioral therapy
- online group CBT-E (Experimental): After randomization, 8-10 patients were assigned to online CBT-E group each time.
  Interventions: Behavioral: online Enhanced Cognitive Behavioral therapy
- waiting group (No Intervention): After randomization, 8-10 patients were assigned to the waiting list each time, and they would be allocated to web-based guided self-help CBT-E or online group CBT-E randomly after a 12-week waiting period.

INTERVENTIONS:
Behavioral: web-based guided self-help Enhanced Cognitive Behavioral therapy — The subjects would learn and practice CBT-E course through the online learning platform for 12 times, and were required to complete the course once a week.
  Arms: web-based guided self-help CBT-E
Behavioral: online Enhanced Cognitive Behavioral therapy — A closed structured group would be established by online video conference for group CBT-E therapy. Each group would receive 12 group sessions, once a week for 120 minutes each time. Each group would be led by two CBT therapists, all of whom are nationally registered psychotherapists with systematic professional training.
  Arms: online group CBT-E

SUMMARY:
Eating disorders with binge eating as the core feature include bulimia nervosa (BN) and binge eating disorder (BED). In recent years, the prevalence rate has increased rapidly, mostly among women, accompanied by emotional problems, physiological complications and increased risks of obesity and depression, which bring great pain to patients. Enhanced Cognitive Behavioral therapy (CBT-E) for eating disorders is an evidence-based and effective first-line psychotherapy for BN and BED. CBT-E is implemented in various forms. In addition to face-to-face therapy, online group CBT-E and guided self-help CBT-E can significantly reduce binge eating in BN and BED patients. However, there are no relevant clinical studies in China. Since 2008, the applicant has carried out CBT treatment and research on eating disorders, translated and published the self-help book "Overcoming Overeating", and accumulated rich clinical research experience. This study intends to establish a set of CBT-E self-help therapy courses suitable for Chinese binge eating patients, and conduct a randomized controlled study of web-based guided self-help CBT-E and online group CBT-E to compare the effectiveness of the treatment modalities in the treatment of binge eating and the feasibility of online guided self-help CBT-E and online group CBT-E in the treatment of binge eating.

ELIGIBILITY:
Inclusion Criteria:

* Han nationality, aged 18-35 years old;
* Students with junior high school education or above;
* Meet the diagnostic criteria of BN or BED in DSM-5, body mass index (BMI)≥18.5 kg/m2;
* no systematic nutritional treatment, psychiatric drug treatment or any form of psychological treatment was received within 1 month before enrollment;
* Each patient must understand the nature of this study and sign informed consent.

Exclusion Criteria:

* Persons meeting other DSM-5 diagnoses other than BN and BED, such as substance abuse/dependence, depression, bipolar disorder, anxiety disorder, obsessive-compulsive disorder, etc., persons at high risk of suicide, persons with strong destructive impulses or antisocial behaviors;
* The patient has severe primary or secondary physical disease or cognitive impairment, which makes the patient unable to complete the required symptom assessment and psychological tests;
* Have received systematic nutritional therapy, individual and group psychotherapy;
* Those who have taken neuroblockers, antidepressants, lithium salts, stimulants, antiepileptics and other psychotropic drugs within the past 1 month;
* Participation in this clinical trial was deemed inappropriate by the investigator for other reasons.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Eating Disorder Examination Questionnaire (EDE-Q) at Post-Treatment and During Follow-Up | Baseline, Week 12 (at the end of treatment), Week 16 (1 month after treatment), week 24 (3 months after treatment)
  Questions 13 to 15 of the Eating Disorder Survey Scale (EDE-Q) were used to assess the proportion of patients with no binge eating behavior in the last 28 days.

SECONDARY OUTCOMES:
Barratt Impulsivity Scale-Version 11 (BIS-11) | Baseline, Week 12 (at the end of treatment), Week 16 (1 month after treatment), week 24 (3 months after treatment)
  To evaluate the changes in impulse suppression ability of patients before and after treatment, the Barratt Impulsivity Scale-11 (BIS-11) comprises 30 questions. Each question is on a 4-point scale from 1 to 4. Scores range from 30 to 120, with higher scores indicating higher levels of impulsivity.
Beck Depression Inventory-Version 2 (BDI-2) | Baseline, Week 12 (at the end of treatment), Week 16 (1 month after treatment), week 24 (3 months after treatment)
  To assess the changes of depressive mood before and after treatment, the Beck Depression Inventory-Version 2 (BDI-2) comprises 21 questions. Each question is on a 4-point scale from 0 to 3. Scores range from 0 to 63, with higher scores indicating higher levels of depression.
Beck Anxiety Inventory (BAI) | Baseline, Week 12 (at the end of treatment), Week 16 (1 month after treatment), week 24 (3 months after treatment)
  To assess the changes of anxiety mood before and after treatment, the Beck Anxiety Inventory (BAI) comprises 21 questions. Each question is on a 4-point scale from 0 to 3. Scores range from 0 to 63, with higher scores indicating higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jue Chen, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and baseline characteristics of participants.
Supporting Information: Study Protocol, SAP
Time Frame: Researchers will share data when the study is completed in December 2024.
Access Criteria: CBT-E; bulimia nervosa; binge eating; online CBT-E

REFERENCES:
- [Background] Agras WS. Cognitive Behavior Therapy for the Eating Disorders. Psychiatr Clin North Am. 2019 Jun;42(2):169-179. doi: 10.1016/j.psc.2019.01.001. Epub 2019 Apr 2. PMID 31046920
- [Background] Hay P, Palavras MA, da Luz FQ, Dos Anjos Garnes S, Sainsbury A, Touyz S, Appolinario JC, Claudino AM. Physical and mental health outcomes of an integrated cognitive behavioural and weight management therapy for people with an eating disorder characterized by binge eating and a high body mass index: a randomized controlled trial. BMC Psychiatry. 2022 May 24;22(1):355. doi: 10.1186/s12888-022-04005-y. PMID 35610603
- [Background] Atwood ME, Friedman A. A systematic review of enhanced cognitive behavioral therapy (CBT-E) for eating disorders. Int J Eat Disord. 2020 Mar;53(3):311-330. doi: 10.1002/eat.23206. Epub 2019 Dec 16. PMID 31840285
- [Background] da Luz FQ, Hay P, Wisniewski L, Cordas T, Sainsbury A. The treatment of binge eating disorder with cognitive behavior therapy and other therapies: An overview and clinical considerations. Obes Rev. 2020 Dec 17. doi: 10.1111/obr.13180. Online ahead of print. PMID 33350574